CLINICAL TRIAL: NCT04386785
Title: Investigator Initiated Safety Study Using the Venclose Vestico (Commercial Name TBD) Radiofrequency (RF) Ablation System for the Treatment of Incompetent Perforator Veins (IPVs)
Brief Title: Venclose RF Ablation System for the Treatment of IPVs
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Venclose, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CL-VAV-001
Record Dates: First submitted 2020-05-07; First posted 2020-05-13 (Actual); Results first posted 2022-05-27 (Actual); Last update posted 2022-05-27 (Actual); Status verified 2022-05

CONDITIONS: Chronic Venous Insufficiency

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- Single-arm: Endovascular thermal ablation in IPV (Experimental)
  Interventions: Device: Radiofrequency (RF) Thermal Ablation of Incompetent Perforator Veins

INTERVENTIONS:
Device: Radiofrequency (RF) Thermal Ablation of Incompetent Perforator Veins — The physician operator will access the IPV and advance the device to the target treatment position using ultrasound guidance. After providing local anesthesia to the vein and surrounding tissues, thermal ablation energy is delivered to the vein wall. After treatment is complete, the device is removed and vessel closure confirmed with duplex ultrasound.

SUMMARY:
A feasibility study conducted in patients with incompetent (i.e. refluxing) perforator veins were treated using the Venclose RF Ablation System.

ELIGIBILITY:
Inclusion Criteria:

* Patient is >= 18 years.
* IPVs to be treated have an outward flow duration of >= 0.5 seconds immediately after release of manual distal compression with patient standing or in Reverse Trendelenburg.
* IPV(s) to be treated have a diameter of ≥ 3.5 mm located caudal edge of ankle.
* Has been diagnosed with refractory symptomatic disease attributable to the IPV to be treated.
* Is able to ambulate.
* Is able to comprehend and has signed the Informed Consent Form (ICF) to participate in the study.
* Is willing and able to comply with the Clinical Investigation Plan and follow-up schedule.

Exclusion Criteria:

* Has venous insufficiency secondary to venous obstruction proximal to the intended treatment site.
* Has thrombus in the vein segment to be treated.
* Has untreated critical limb ischemia from peripheral arterial disease.
* Is undergoing active anticoagulant therapy for Deep Vein Thrombosis or other conditions (e.g., warfarin, direct oral anticoagulant or low molecular weight heparin) or has a history of Deep Vein Thrombosis within the last 6 months or hypercoagulable state.
* Patients with known bleeding or clotting disorders or unwilling or unable to frequently ambulate post-operatively.
* Has had prior venous procedures in the study limb within the last 30 days (including thrombolysis, thrombectomy, stenting, ablation, phlebectomy, visual or foam sclerotherapy).
* Has undergone or is expected to undergo any major surgery within 30 days prior to or following the study procedure.
* Has a condition, judged by the treating physician, that may jeopardize the patient's well-being and/or confound the results or the soundness of the study.
* Is pregnant or lactating at the time of the study procedure or is intending on becoming pregnant within 30 days following the study procedure.
* Is participating in another clinical study that is contraindicated to the treatment or outcomes of this investigation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2020-05-23 (Actual); Primary Completion 2021-04-13 (Actual); Study Completion 2021-05-13 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey Carr, MD, Principal Investigator — Vein Center of East Texas at CardioStream
Locations (1):
- Vein Center of East Texas at CardioStream, Tyler, Texas, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Units Other Than Participants: Incompetent Perforator Veins
Period: Overall Study
Arm/Group | Single-arm: Endovascular Thermal Ablation in IPV
Started | 27; 30 Incompetent Perforator Veins
Completed | 27; 30 Incompetent Perforator Veins
Not Completed | 0; 0 Incompetent Perforator Veins

BASELINE CHARACTERISTICS:
Units Other Than Participants: IPVs
Arm/Group | Single-arm: Endovascular Thermal Ablation in IPV
Number analyzed (Participants) | 27
Number analyzed (IPVs) | 30
Age, Continuous [Mean (Standard Deviation); unit: years] | 67.8 (14.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11
  Male | 16
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
  Participants
    number analyzed (Participants) | 0
Region of Enrollment [Number; unit: participants]
  United States | 27
Weight [Mean (Standard Deviation); unit: pounds] | 235.2 (53.6)
Height [Mean (Standard Deviation); unit: inches] | 66.7 (18.5)
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m^2] | 37.1 (7.9)
Number of Veins [Count of Units; unit: IPVs]
  Female | 14
  Male | 16
CEAP Classification [Count of Units; unit: IPVs] — Status of clinical signs and symptoms of lower limb venous disease as measured by the physician using the Clinical Etiologic Anatomic Pathophysiologic (CEAP) system.
  C0: No visible or palpable signs of venous disease C1: Telangiectasias or reticular veins C2: Varicose veins C3: Edema C4: Changes in skin and subcutaneous tissue secondary C5: Healed C6: Active venous ulcer
  IPVs
    C0 | 0
    C1 | 0
    C2 | 0
    C3 | 0
    C4 | 13
    C5 | 7
    C6 | 10

OUTCOME MEASURES:

1. Primary Outcome: Safety: AEs, SAEs, ADEs, SADEs, UADEs
Description: Procedure related adverse events (AE), serious adverse events (SAE), adverse device effects (ADE), serious adverse device effects (SADE) and unanticipated adverse device effects (UADE) will be monitored analyzed for acceptability post study.
Time Frame: 3-day post-procedure
Measure: Number; unit: Events
Arm/Group | Single-arm: Endovascular Thermal Ablation in IPV
Number analyzed (Participants) | 27
Events
  Procedure related AEs | 0
  Procedure related SAEs | 0
  ADEs | 0
  SADEs | 0
  UADEs | 0

2. Primary Outcome: Safety: AEs, SAEs, ADEs, SADEs, UADEs
Description: as for outcome 1
Time Frame: 15-day post-procedure
Measure: Number; unit: Events
Arm/Group | Single-arm: Endovascular Thermal Ablation in IPV
Number analyzed (Participants) | 27
Events
  Procedure related AEs | 0
  Procedure related SAEs | 0
  ADEs | 0
  SADEs | 0
  UADEs | 0

3. Primary Outcome: Safety: AEs, SAEs, ADEs, SADEs, UADEs
Description: as for outcome 1
Time Frame: 30-day post-procedure
Measure: Number; unit: Events
Arm/Group | Single-arm: Endovascular Thermal Ablation in IPV
Number analyzed (Participants) | 27
Events
  Procedure related AEs | 0
  Procedure related SAEs | 0
  ADEs | 0
  SADEs | 0
  UADEs | 0

4. Primary Outcome: Effectiveness: Technical Success
Description: Technical success defined as successful access and entry into the IPV to be ablated and the ability to deliver the intended energy to the target vein segment, will be evaluated.
Time Frame: Day of procedure
Measure: Count of Units; unit: IPVs
Units Other Than Participants: IPVs
Arm/Group | Single-arm: Endovascular Thermal Ablation in IPV
Number analyzed (Participants) | 27
Number analyzed (IPVs) | 30
IPVs | 30

5. Primary Outcome: Effectiveness: Successful Access and Entry Into the IPV
Description: as for outcome 4
Time Frame: 3-day post ablation
Measure: Count of Units; unit: IPVs
Units Other Than Participants: IPVs
Arm/Group | Single-arm: Endovascular Thermal Ablation in IPV
Number analyzed (Participants) | 27
Number analyzed (IPVs) | 30
IPVs | 30

6. Primary Outcome: Effectiveness: Technical Success
Description: as for outcome 4
Time Frame: 15-day post ablation
Measure: Count of Units; unit: IPVs
Units Other Than Participants: IPVs
Arm/Group | Single-arm: Endovascular Thermal Ablation in IPV
Number analyzed (Participants) | 27
Number analyzed (IPVs) | 30
IPVs | 30

7. Primary Outcome: Effectiveness: Technical Success
Description: as for outcome 4
Time Frame: 30-day post ablation
Measure: Count of Units; unit: IPVs
Units Other Than Participants: IPVs
Arm/Group | Single-arm: Endovascular Thermal Ablation in IPV
Number analyzed (Participants) | 27
Number analyzed (IPVs) | 30
IPVs | 30

8. Secondary Outcome: Acute Ablation Success
Description: The acute ablation success endpoint is defined as complete lack of flow or IPV disappearance in the treated segment (vessel occlusion). Success will be measured by Duplex Ultrasound imaging post-procedure.
Time Frame: 3-day post-procedure follow-up
Measure: Count of Units; unit: IPVs
Units Other Than Participants: IPVs
Arm/Group | Single-arm: Endovascular Thermal Ablation in IPV
Number analyzed (Participants) | 27
Number analyzed (IPVs) | 30
IPVs | 23

9. Secondary Outcome: Acute Ablation Success
Description: as for outcome 8
Time Frame: 15-day post-procedure
Measure: Count of Units; unit: IPVs
Units Other Than Participants: IPVs
Arm/Group | Single-arm: Endovascular Thermal Ablation in IPV
Number analyzed (Participants) | 27
Number analyzed (IPVs) | 30
IPVs | 22

10. Secondary Outcome: Acute Ablation Success
Description: as for outcome 8
Time Frame: 30-day post-procedure
Measure: Count of Units; unit: IPVs
Units Other Than Participants: IPVs
Arm/Group | Single-arm: Endovascular Thermal Ablation in IPV
Number analyzed (Participants) | 27
Number analyzed (IPVs) | 30
IPVs | 24

11. Secondary Outcome: Reflux
Description: Presence of reflux in the treated IPV will be recorded at each time point and an overall absence of reflux rate (i.e. reflux free rate) will be documented at each follow-up time point.
Time Frame: 3-day post-procedure
Measure: Count of Units; unit: IPVs
Units Other Than Participants: IPVs
Arm/Group | Single-arm: Endovascular Thermal Ablation in IPV
Number analyzed (Participants) | 27
Number analyzed (IPVs) | 30
IPVs | 26

12. Secondary Outcome: Reflux
Description: as for outcome 11
Time Frame: 15-day post-procedure
Measure: Count of Units; unit: IPVs
Units Other Than Participants: IPVs
Arm/Group | Single-arm: Endovascular Thermal Ablation in IPV
Number analyzed (Participants) | 27
Number analyzed (IPVs) | 30
IPVs | 25

13. Secondary Outcome: Reflux
Description: as for outcome 11
Time Frame: 30-day post-procedure
Measure: Count of Units; unit: IPVs
Units Other Than Participants: IPVs
Arm/Group | Single-arm: Endovascular Thermal Ablation in IPV
Number analyzed (Participants) | 27
Number analyzed (IPVs) | 30
IPVs | 28

ADVERSE EVENTS:
Time Frame: AEs, SAEs, ADEs, SADEs, UADEs were captured for each participant at Baseline, Day of Procedure, and then 3-day, 15-day, and 30-day post-procedure follow-up visits.
Arm/Group | Single-arm: Endovascular Thermal Ablation in IPV
All-Cause Mortality (participants affected / at risk) | 0/27
Serious Adverse Events (participants affected / at risk) | 0/27
Other Adverse Events (participants affected / at risk) | 0/27

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2020-04-14): https://cdn.clinicaltrials.gov/large-docs/85/NCT04386785/Prot_SAP_000.pdf
  • Informed Consent Form (2020-04-14): https://cdn.clinicaltrials.gov/large-docs/85/NCT04386785/ICF_001.pdf